CLINICAL TRIAL: NCT07028268
Title: A Multicenter, Randomized, Double-Blind, Positively Controlled Phase II Clinical Study Evaluating the Efficacy and Safety of SHR-2017 Injection in Patients With Bone Metastases From Solid Tumors
Brief Title: A Trial of SHR-2017 Injection in Patients With Bone Metastases From Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-2017-201
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-06

CONDITIONS: For Prevention of Bone Events in Patients With Bone Metastases From Solid Tumors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group A: SHR-2017、Denosumab placebo (Experimental)
  Interventions: Drug: SHR-2017、Denosumab placebo
- Treatment group B: SHR-2017、Denosumab placebo (Experimental)
  Interventions: Drug: SHR-2017、Denosumab placebo
- Treatment group C: Denosumab；SHR-2017 placebo (Active Comparator)
  Interventions: Drug: Denosumab；SHR-2017 placebo

INTERVENTIONS:
Drug: SHR-2017、Denosumab placebo — SHR-2017; high dose ；Denosumab placebo
  Arms: Treatment group A: SHR-2017、Denosumab placebo
Drug: SHR-2017、Denosumab placebo — SHR-2017; low dose ；Denosumab placebo
  Arms: Treatment group B: SHR-2017、Denosumab placebo
Drug: Denosumab；SHR-2017 placebo — Denosumab；SHR-2017 placebo
  Arms: Treatment group C: Denosumab；SHR-2017 placebo

SUMMARY:
The study is being conducted to evaluate the efficacy, and safety of SHR-2017 Injection in Patients with Bone Metastases from Solid Tumors. To explore the reasonable dosage of SHR-2017 Injection for Bone Metastases from Solid Tumors

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent；
2. Male or female, ≥18 years of age；
3. Histologically or cytologically confirmed solid tumors；
4. At least 1 bone metastasis demonstrated by radiologic imaging or histopathology；
5. Eastern Cooperative Oncology Group performance Status≤2。
6. Life expectancy was judged by the investigators to be at least 6 months;
7. Adequate organ function at Screening
8. Female subjects with a negative blood pregnancy test and are not breastfeeding

Exclusion Criteria:

1. Pre-existing or comorbid related oral diseases or oral cavity requiring surgery, etc；
2. History of major joint (e.g., hip, knee, or shoulder) trauma or surgery prior to the first dose of the drug；
3. Received radiotherapeutic drugs or bone radiotherapy prior to the first study drug administration
4. Any cardiovascular disease for which the investigator considers the subject unfit to participate in the study
5. resting tachycardia or resting bradycardia;
6. The subject's pain is predominantly from pain unrelated to the bone metastases;
7. Subject is unable to perform a pain assessment;
8. Symptomatic or treatment-requiring brain metastases or other central nervous system metastases
9. Comorbid infectious disease
10. Prior receipt of exogenous nerve growth factor or anti-nerve growth factor antibodies;
11. Prior history of allergy to relevant drug ingredients or components;
12. Participation in other clinical trials within a certain period of time
13. Subjects who, in the opinion of the investigator, have any other factors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Time to pain relief | randomization to 48 weeks after administration
  Analgesic evaluation using NRS scores
percentage of change in the bone turnover marker urine N-telopeptide corrected for urine creatinine (uNTx/Cr) from baseline to study week 13 | randomization to 13 weeks after administration

SECONDARY OUTCOMES:
Time to first on-study SRE (defined as pathologic fracture, radiation or surgery to bone, or spinalcord compression). | randomization to 72 weeks after administration
Change from Baseline in the daily average pain intensity in the index bonemetastasis cancer pain site. | randomization to 48 weeks after administration
Change from Baseline in the daily worst pain intensity in the index bonemetastasis cancer pain site. | randomization to 48 weeks after administration
Response as defined by a ≥2 point reduction from Baseline in the daily average and daily worst pain intensity NRS score in the index bone metastasis cancer pain site | randomization to 48 weeks after administration
Average daily total opioid consumption (in mg of morphine equivalent doses) | randomization to 48 weeks after administration

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided